CLINICAL TRIAL: NCT04394390
Title: Vitamin D Levels in SARS-CoV-2: Do Current Adequacy Thresholds Reflect Clinical Risk? Insights From a Large Turkish Cohort
Status: Completed | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Taner Dandinoğlu, Taner Dandinoglu MD. Principal Investigator, Physical Medicine and Rehabilitation (PMR) specialist., Bursa City Hospital
Other Study IDs: 2020-PMR-1
Record Dates: First submitted 2020-05-18; First posted 2020-05-19 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: COVID; Vitamin D Deficiency
Keywords: covid-19, infection, vitamin D, prevention
MeSH Terms: conditions — Vitamin D Deficiency; COVID-19; Infections | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: vitamin d — vitamin D levels
  Other Names: vitamin D levels

SUMMARY:
Blood vitamin D levels may be associated with severity of viral infections. To find out If there is a statistically significant relation between blood 25-hydroxy vitamin D (25(OH)D) levels and disease severity, patients with Covid-19 viral infection were investigated.

DETAILED DESCRIPTION:
Purpose:

Vitamin D a steroid hormone has profound effects on human immunity. Active vitamin D, 1,25(OH)2D acts as an immune system modulator, preventing excessive expression of inflammatory cytokines and increasing the 'oxidative burst' potential of macrophages. Epidemiological data has linked vitamin D deficiency to increased susceptibility to acute viral respiratory infections.

There is evidence that some patients with severe COVID-19 experience a cytokine storm with production of large quantities of interleukins, specifically IL-1 and IL-6. Moreover it was hipotiesied that the sufficient vitamin D levels may help to decrease IL-6 levels like tocizulamab which is a potent blocking agent of the IL-6 receptor.

In this observational study, possible relation between the disease and vitamin D levels were investigated in COVİD-19 patients.

Material and Methods:

To find out vitamin D levels and it's relation with the disease severity serum 25-hydroxy-vitamin D levels will be measured in nearly 1100 confirmed COVİD-19 patients. Same patients will also be evaluated for vital signs, laboratory and pulmoner CT findings. Demographic and medical data will also be collected. Statically significant positive or negative results and the comparison of these findings will be presented.

Presenting blood vitamin- D levels and it's possible assosiation with disease severity may inspire new perspectives for future trials spesifically focusing vitamin D levels.

ELIGIBILITY:
To find out vitamin D levels and it's relation with the disease severity serum 25-hydroxy-vitamin D levels, 1100 confirmed Covid-19 patients with available laboratory findings were included.

Exlucion Criterias:

Using immunsuppresan medical treatment. Using vitamin D or replacement history of vitamin D in last 3 months. Patients with malnutrition, immun deficiency, chronic infections, chronic other diseases such as rheumatoid arthritis, ankylosing spondilitis, lupus, hemplegia, paraplegia etc.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1100 confirmed COVİD-19 patients (PCR)
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
laboratory measured vitamin D levels | 12 months
  serum 25-hydroxy-vitamin D levels

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa City Hospital, Bursa, Dogankoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Research data will be available upon request from authors
  (Taner Dandinoglu MD. e-mail: dandinoglu@gmail.com, Sinem Akselim MD e-mail: sinemakselim@gmail.com)

REFERENCES:
- [Background] Jayawardena R, Sooriyaarachchi P, Chourdakis M, Jeewandara C, Ranasinghe P. Enhancing immunity in viral infections, with special emphasis on COVID-19: A review. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):367-382. doi: 10.1016/j.dsx.2020.04.015. Epub 2020 Apr 16. PMID 32334392
- [Background] Silberstein M. Vitamin D: A simpler alternative to tocilizumab for trial in COVID-19? Med Hypotheses. 2020 Jul;140:109767. doi: 10.1016/j.mehy.2020.109767. Epub 2020 Apr 23. PMID 32353742